CLINICAL TRIAL: NCT01447927
Title: Randomized Double Blind Placebo Controlled Trial of Barrett's Esophagus Chemoprevention With Metformin
Brief Title: Metformin Hydrochloride in Preventing Esophageal Cancer in Patients With Barrett Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2011-03451; MAY10-15-03; MAYO-MAY10-15-03; CDR0000698069
Record Dates: First submitted 2011-10-05; First posted 2011-10-06 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Barrett Esophagus; Esophageal Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Patients receive extended-release metformin hydrochloride PO QD on week 1, and BID on weeks 2-12 (QAM QPM on week 3) in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: metformin hydrochloride
- Arm II (Placebo Comparator): Patients receive extended-release placebo PO QD on week 1and BID on weeks 2-12 (QAM and QPM on week 3) in the absence of unacceptable toxicity or disease progression.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO QD and BID
  Other Names: Glucophage
  Arms: Arm I
Other: placebo — Given PO QD and BID
  Other Names: PLCB
  Arms: Arm II

SUMMARY:
This randomized phase II trial studies how well metformin hydrochloride works in preventing esophageal cancer in patients with Barrett esophagus. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of metformin hydrochloride may keep esophageal cancer from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the percent change in the mean pS6K1 immunostaining from baseline in mucosal Barrett esophagus (BE) biopsies among patients assigned to 2,000 mg metformin hydrochloride once daily (QD) versus placebo as determined from Barrett mucosal biopsy samples obtained pre- and post-intervention.

SECONDARY OBJECTIVES:

I. To evaluate adverse events associated with the two intervention arms.

TERTIARY OBJECTIVES:

I. To assess the effects of metformin hydrochloride 2,000 mg QD versus placebo on the changes in pS6K1 using traditional IHC categories.

II. To assess the effects of metformin hydrochloride 2,000 mg QD versus placebo on absolute change in pS6K1.

III. To assess changes in serum markers (metformin hydrochloride, fasting insulin, HOMA-IR, IGF-1, IGF-2, IGFBP-1, IGFBP-3, fasting leptin, and fasting adiponectin) as determined from serum samples obtained pre- and post-intervention.

IV. To assess changes in proliferation (Ki-67) and apoptosis (cleaved caspase 3) as determined from Barrett mucosal biopsy samples obtained pre- and post-intervention.

V. To assess changes in molecular mediators of the insulin pathway (p-IRS-1, p-AKT^Serine 473) as determined from Barrett mucosal biopsy samples obtained pre- and post-intervention.

VI. To assess changes in relative activity of AMPK (phosphorylated AMPK/total AMPK ratio) and molecular mediators of AMP kinase (p-mTOR, pS6K1^Serine 235) as determined from Barrett mucosal biopsy samples obtained pre- and post-intervention.

VII. To assess changes in Programmed Cell Death 4 expression and miR-21 as determined from Barrett mucosal biopsy samples pre- and post-intervention.

VIII. To establish a biospecimen repository archive for future correlative studies.

OUTLINE: This is a multicenter study.

Patients are stratified according to nonsteroidal anti-inflammatory drugs use (regular vs no regular), body mass index (≥ 30 kg/m² vs < 30 kg/m²), gender (male vs female), and length of Barrett (2.00 to 4.99 cm vs ≥ 5.00 cm). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive extended-release metformin hydrochloride orally (PO) once daily (QD) on week 1, and twice daily (BID) on weeks 2-12 (every morning [QAM] and every evening [QPM] on week 3) in the absence of unacceptable toxicity or disease progression.

Arm II: Patients receive extended-release placebo PO QD on week 1 and BID on weeks 2-12 (QAM and QPM on week 3) in the absence of unacceptable toxicity or disease progression.

Blood, tissue, and mucosal tissue samples are collected at baseline and after completion of study treatment for pS6K1 analysis and other serum, mucosal, and molecular markers studies by IHC, ELISA, western blotting, and high-performance liquid chromatography (HPLC) methods.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Barrett esophagus, with no dysplasia, indeterminate for dysplasia, or low-grade dysplasia as defined by the presence of specialized columnar epithelium on histology and >= 2 cm of involvement on endoscopy
* Adequate Barrett mucosa, which is defined as >= 1 out of 4 research samples (i.e., >= 25%) with >= 50% intestinal metaplasia in biopsies required to satisfy the endpoints of the study
* No history of esophageal carcinoma or other cancer(s) (except for non-melanoma skin cancers)
* No erosive esophagitis or ulcerative esophagitis, unless treatment with a proton pump inhibitor (PPI) results in healed erosions or ulcers prior to entry endoscopy
* No history of high-grade dysplasia or cancer (confirmed locally by esophagogastroduodenoscopy [EGD] and Pathology reports)

  * No ulcer, plaque, nodule, stricture, or other luminal irregularity within the Barrett segment, unless clinical biopsy produces no evidence of high-grade dysplasia or cancer
* ECOG performance status =< 1
* Hemoglobin >= 10 g/dL
* Leukocytes >= 3,000/mL (>= 2,500/mL for African-American participants)
* Absolute neutrophil count >= 1,500/mL (>= 1,000/mL for African-American participants)
* Platelets >= 100,000/mL
* Total bilirubin =< institutional upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) =< 1.5 times institutional ULN
* Creatinine =< institutional ULN
* Willingness to provide tissue samples for research purposes
* No contraindication to esophagogastroduodenoscopy (EGD)
* Willingness, for both men and women, to use adequate contraception (hormonal or barrier method of birth control; surgical intervention; abstinence) prior to study entry and for the duration of study participation
* A negative (serum or urine) pregnancy test done =< 7 days prior to Pre-Registration, for women of childbearing potential only
* No pregnant or nursing women
* No participants with diabetes mellitus
* No history of vitamin B12 deficiency or megaloblastic anemia
* No history of lactic acidosis
* No diseases associated with weight loss: anorexia, bulimia, or nausea
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin
* No participants with HIV, cirrhosis of any cause, NASH (non-alcoholic steatohepatitis), or hepatitis (auto-immune or infectious)

  * For participants diagnosed with any other hepatic impairment, consult with protocol principal investigator (PI)
* No metabolic acidosis, acute or chronic, including ketoacidosis
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; this includes significant medical conditions including renal failure, hepatic failure, sepsis, and hypoxia
* No genetics disorders such as family history of hereditary gastrointestinal polyp disorder (e.g., familial adenomatous polyposis [FAP], hereditary non-polyposis colorectal cancer [HNPCC], Peutz-Jegher disease)
* No chronic alcohol use or a history of alcohol abuse (defined as ingestion of >= 3 drinks per day)
* No kidney disease or renal insufficiency (defined as serum creatinine outside the normal institutional limits)
* Currently on a proton pump inhibitor (PPI) >= 4 weeks (any PPI taken at least once daily is acceptable)
* No medication(s) for weight loss ≤ 2 months prior to Pre-Registration
* No treatment with medications that may increase metformin hydrochloride levels: cationic drugs, e.g., digoxin, amiloride, procainamide, ranitidine, trimethoprim, quinidine, quinine, vancomycin, triamterene, and morphine
* No treatment with other oral hypoglycemic agents
* No participant use of metformin, cimetidine (Tagamet), furosemide (Lasix), or nifedipine (Cardizem), or any other drug contraindicated for use with metformin
* No receipt of any other investigational agents =< 3 months prior to Pre-Registration, except innocuous agents with no known interaction with the study agent (e.g., standard dose multivitamins or topical agents for limited skin conditions), at the discretion of the Protocol Lead Investigator at each Participating Site
* No participants who have undergone ablation or other local therapies (e.g., percutaneous dilatational tracheostomy [PDT], cryotherapy, radiofrequency, argon plasma coagulation [APC], or multipolar electrocoagulation [MPEC])

  * Patients treated with endoscopic mucosal resection [EMR] allowed
* No participants anticipating elective surgery during the study period
* No participants planning to undergo elective radiologic studies involving intravascular administration of iodinated contrast materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Chak, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (7):
- United States (5):
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center - Shadyside Hospital, Pittsburgh, Pennsylvania
- University of Toronto, Toronto, Ontario, Canada
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Chak A, Buttar NS, Foster NR, Seisler DK, Marcon NE, Schoen R, Cruz-Correa MR, Falk GW, Sharma P, Hur C, Katzka DA, Rodriguez LM, Richmond E, Sharma AN, Smyrk TC, Mandrekar SJ, Limburg PJ; Cancer Prevention Network. Metformin does not reduce markers of cell proliferation in esophageal tissues of patients with Barrett's esophagus. Clin Gastroenterol Hepatol. 2015 Apr;13(4):665-72.e1-4. doi: 10.1016/j.cgh.2014.08.040. Epub 2014 Sep 15. PMID 25218668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-three subjects were pre-registered through 12 Cancer Prevention Network (CPN) member organizations from February 2012 and January 2013.
Pre-assignment Details: One subject withdrew post-randomization and did not receive any treatment and 18 subjects were excluded from the trial before assignment to groups: 8 out of range lab values, 4 high grade dysplasia/esophagitis/esophageal stricture, 2 intestinal metaplasia on <25% of biopsies, and 4 other reasons.
Groups:
- Metformin: Patients receive extended-release metformin hydrochloride orally (PO) once daily (QD) on week 1, and twice daily (BID) on weeks 2-12 (every morning (QAM) every evening (QPM) on week 3) in the absence of unacceptable toxicity or disease progression.
- Placebo: Patients receive extended-release placebo orally (PO) once daily (QD) on week 1and BID on weeks 2-12 (every morning (QAM) and every evening (QPM) on week 3) in the absence of unacceptable toxicity or disease progression.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 38 | 36
Completed | 33 | 33
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin: Patients receive extended-release metformin hydrochloride PO QD on week 1, and BID on weeks 2-12 (QAM QPM on week 3) in the absence of unacceptable toxicity or disease progression.
- Placebo: Patients receive extended-release placebo PO QD on week 1and BID on weeks 2-12 (QAM and QPM on week 3) in the absence of unacceptable toxicity or disease progression.
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Median (Full Range); unit: years] | 60.5 [20.0 to 81.0] | 60.5 [39.0 to 79.0] | 60.5 [20.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 30 | 28 | 58
Performance Score [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0-Fully active | 37 | 35 | 72
    1-Ambulatory, restricted strenuous activity | 1 | 1 | 2
Body Mass Index [Median (Full Range); unit: kg/m^2] | 30.1 [22.3 to 44.5] | 29.9 [20.2 to 52.0] | 30.0 [20.2 to 52.0]
Length of Barrett's segment [Number; unit: participants]
  <5 cm of circumferential involvement | 11 | 11 | 22
  >=5 cm of circumferential involvement | 27 | 25 | 52
Non-steroidal anti-inflammatory drug (NSAID) use [Number; unit: participants]
  Regular Use | 9 | 8 | 17
  No Regular Use | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Median pS6K1 Immunostaining Among Participants With Barrett Esophagus
Description: The percent change in pS6K1 was calculated as month 3 pS6k1 values minus baseline pS6k1 values, then divide by baseline pS6k1 values and multiply by 100.
Time Frame: Baseline to 3 months
Population: Participants were considered evaluable for primary endpoint if pS6K1 data were available from both the pre- and post-intervention evaluations based on the intent-to-treat principle.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 36 | 33
percentage of change | 1.4 (157.1) [-88.1 to 694.0] | -14.7 (301.0) [-97.7 to 1646.1]
Statistical Analysis 1: Comparison: Metformin vs Placebo; The null hypothesis was that the percent change in mean pS6K1 values (from pre to post) was the same or increased for the metformin arm as compared to placebo. Assuming equal standard deviations (i.e. 50%) across the metformin and placebo groups, 30 participants per arm yielded 84% power to detect at least a 35% decrease in the metformin arm as compared to placebo, using a 1-sided t-test with a significant level of 0.05; Test type: Superiority or Other; p = 0.7981, Wilcoxon Rank-Rum Test (1-sided)

2. Secondary Outcome: Overall Adverse Event Rates
Description: Number of patients that experienced adverse events (grade 1 or above) as measured by NCI CTCAE (Common Terminology Criteria for Adverse Events) v. 4.0.
  The data reported in the table include only the commonly occurring adverse events (3 or more events).
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 38 | 36
participants
  Abdominal Pain | 6 | 0
  Cough | 0 | 3
  Diarrhea | 10 | 5
  Dyspepsia | 2 | 3
  Fatigue | 4 | 1
  Flatulence | 2 | 2
  Flu like symptoms | 1 | 2
  Gastrointestinal disorders - other, specify | 2 | 2
  Headache | 3 | 2
  Nausea | 5 | 3

ADVERSE EVENTS:
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/38
Other Adverse Events (participants affected / at risk) | 23/36 | 26/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Metformin (N=38)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Metformin (N=38)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 10 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (4)
Flu like symptoms (General disorders) | 2 (2) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less